CLINICAL TRIAL: NCT00512759
Title: Goal-Directed Afterload Reduction in Acute Congestive Cardiac Decompensation Study (GALACTIC)
Brief Title: Goal-directed Afterload Reduction in Acute Congestive Cardiac Decompensation Study
Acronym: GALACTIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Christian Müller, MD, Prof. Dr. med., University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GALACTIC
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Acute Heart Failure
MeSH Terms: interventions — Ramipril; candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care (No Intervention): Standard of care of acute decompensated heart failure will be according to the current guidelines of the European Society of Cardiology (ESC).
- Intervention (Experimental): Early goal-directed preload and afterload decrement using a fixed therapy schedule including sublingual or nitrospray and transdermal nitrates together with hydralazine, followed by rapid up-titration of ACE-inhibitors , AT-receptor blockers or neprilysin inhibitors/AT-receptor blockers to achieve maximal vasodilatation with a target systolic blood pressure of 90-110 mmHg. All other elements of treatment will be according to the current guidelines of the European Society of Cardiology (ESC)
  Interventions: Drug: Goal-directed preload and afterload decrement

INTERVENTIONS:
Drug: Goal-directed preload and afterload decrement — Early goal-directed preload and afterload decrement with a target systolic blood pressure (RR) of 90-110 mmHg for the entire hospitalization using sublingual nitrates (Nitroglycerin Streuli®) or nitrospray (Corangin Nitrospray®) transdermal nitrates (Nitroderm TTS 10®), ACE-inhibitors (Triatec®) and/or ARB (Atacand®).
  Other Names: Nitroglycerin Streuli®; Nitroderm TTS 10®; Triatec®; Atacand®; Corangin Nitrospray®
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine whether an early goal-directed decrement of preload and afterload with a target systolic blood pressure of 90-110 mmHg by aggressive vasodilatation in patients with acute HF in the non-ICU setting is safe, and leads to a better clinical and economical outcome

DETAILED DESCRIPTION:
Background: Heart failure (HF) is a chronic and progressive illness resulting from a variety of cardiac causes, including ischemic and valvular heart disease, dilatative cardiomyopathy or hypertension. HF may also develop suddenly, particularly as a complication of acute myocardial infarction or as an acute exacerbation in patients with previously compensated chronic HF. Acute HF requires immediate treatment that centers on reducing myocardial oxygen demand and augmenting forward blood flow by removal of excess fluid with diuretics and reduction of preload and afterload with vasodilatators. The aging of our population and the higher number of patients surviving acute myocardial infarctions have lead to a dramatic increase in the incidence and prevalence of HF, and obviously also on total cost burden of the disease. For multiple reasons including need for restrictive use of the limited number of ICU hospital beds the vast majority of elderly patients with acute HF are treated in a non-ICU setting. Unfortunately, the optimal treatment of acute HF in the non-ICU setting is not well defined. Pathophysiological considerations and preliminary data from the ICU setting suggest that aggressive venous and arterial vasodilation may improve short and long-term outcome.

Aim: To test the hypotheses that:

• An early goal-directed decrement of preload and afterload with a target systolic blood pressure of 90-110 mmHg by aggressive vasodilatation in patients with acute HF in the non-ICU setting is safe, and leads to a better clinical and economical outcome

Methods:

Design: Prospective, randomized, controlled, open label, interventional study Setting: University Hospital Basel Patients: Patients with acute HF not requiring ICU admission

Patients admitted to the emergency department with acute HF will be randomized to:

* Early goal-directed preload and afterload decrement using a fixed therapy schedule including sublingual and transdermal nitrates, and hydralazine, followed by rapid up-titration of ACE-inhibitors or AT-receptor blockers to achieve maximal vasodilatation with a target systolic blood pressure of 90-110 mmHg. All other elements of treatment will be according to the current guidelines of the European Society of Cardiology (ESC)
* Standard treatment of acute HF according to the current guidelines of the ESC.

Clinical Significance: Despite the clinical and economical importance of acute HF, the optimal treatment of acute HF is ill-defined. We strongly believe that our novel therapeutic strategy will significantly reduce morbidity, length of hospitalisation, and possibly mortality of affected patients. This would represent a first major step for an evidence-based management of this common condition. Documenting medical and economic benefit of a simple, safe, and inexpensive medical therapy in a randomised controlled clinical trial would provide evidence-based care for the majority of patients presenting with acute HF worldwide. All drugs applied in our strategy are off-patent and therefore relatively low-cost. Successful implication of our treatment algorithm has the potential to significantly reduce treatment costs.

ELIGIBILITY:
Inclusion Criteria:

* Acute HF expressed by acute dyspnea New York Heart Association (NYHA) class III or IV, and a BNP-level ≥ 500 pg/ml. The diagnosis of acute HF is additionally based on typical symptoms and clinical findings, supported by appropriate investigations such as ECG, chest X-ray, and Doppler-echocardiography as recommended by current ESC guidelines on the diagnosis and treatment of acute HF

Exclusion Criteria:

* Cardiopulmonary resuscitation < 7 days
* Cardiogenic shock, ST-elevation myocardial infarction, or other clinical conditions that require immediate ICU admission or urgent PTCA
* Systolic blood pressure lower than 100 mmHg at presentation
* Primary rhythmogenic cause of acute decompensation (ventricular tachycardia, reentry tachycardia, atrial fibrillation or atrial flutter with a ventricular rate exceeding 140 beats per minute)
* NSTEMI as primary diagnosis
* Severe aortic stenosis
* Adult congenital heart disease as primary cause of acute HF
* Hypertrophic obstructive cardiomyopathy
* Chronic kidney disease with creatinin levels > 250 µmol/l
* Bilateral renal artery stenosis
* Severe sepsis or other causes of high output failure
* Cirrhosis of the liver CHILD class C
* Previous adverse reactions to nitrates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 781 (Actual)
Dates: Start 2007-12-10 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
Death or re-hospitalization from HF | 180 days
  Death or re-hospitalization due to heart failure at 180 days

SECONDARY OUTCOMES:
All-cause mortality | 180 days
  All-cause mortality at 180 days
HF re-hospitalization | 180 days
  Re-hospitalization due to heart failure at 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mueller, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (12):
- Hospital Sao Paolo, São Paulo, Brazil
- Bulgaria (3):
  - 5-th Multifunctional Hospital for Active Treatment, Sofia
  - National Transport Hospital "Tsar Boris III", Sofia
  - University Hospital "Tsaritsa Joanna-ISUL", Sofia
- Germany (2):
  - University Hospital Mainz, Mainz
  - Nuremberg Hospital, Nuremberg
- Spain (2):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
- Switzerland (4):
  - University Hospital Basel, Basel, Canton of Basel-City
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Luzern, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen

REFERENCES:
- [Derived] Wussler D, Belkin M, Maeder MT, Walter J, Shrestha S, Kupska K, Stierli M, Flores D, Kozhuharov N, Gualandro DM, de Oliveira Junior MT, Sabti Z, Noveanu M, Socrates T, Bayes-Genis A, Sionis A, Simon P, Michou E, Gujer S, Gori T, Wenzel P, Pfister O, Arenja N, Kobza R, Rickli H, Breidthardt T, Munzel T, Mueller C; GALACTIC Investigators. Comprehensive vasodilatation in women with acute heart failure: Novel insights from the GALACTIC randomized controlled trial. Eur J Heart Fail. 2023 Dec;25(12):2218-2229. doi: 10.1002/ejhf.3065. Epub 2023 Nov 9. PMID 37871997
- [Derived] Kozhuharov N, Goudev A, Flores D, Maeder MT, Walter J, Shrestha S, Gualandro DM, de Oliveira Junior MT, Sabti Z, Muller B, Noveanu M, Socrates T, Ziller R, Bayes-Genis A, Sionis A, Simon P, Michou E, Gujer S, Gori T, Wenzel P, Pfister O, Conen D, Kapos I, Kobza R, Rickli H, Breidthardt T, Munzel T, Erne P, Mueller C; GALACTIC Investigators; Mueller C, Erne P, Muller B, Rickli H, Maeder M, Tavares de Oliveira M Jr, Munzel T, Bayes-Genis A, Sionis A, Goudev A, Dimov B, Hartwiger S, Arenja N, Glatz B, Herr N, Isenrich R, Mosimann T, Twerenbold R, Boeddinghaus J, Nestelberger T, Puelacher C, Freese M, Vogele J, Meissner K, Martin J, Strebel I, Wussler D, Schumacher C, Osswald S, Vogt F, Hilti J, Barata S, Schneider D, Schwarz J, Fitze B, Hartwiger S, Arenja N, Glatz B, Herr N, Isenrich R, Mosimann T, Twerenbold R, Boeddinghaus J, Nestelberger T, Puelacher C, Freese M, Vogele J, Meissner K, Martin J, Strebel I, Wussler D, Schumacher C, Osswald S, Vogt F, Hilti J, Barata S, Schneider D, Schwarz J, Fitze B, Arenja N, Rentsch K, Bossa A, Jallad S, Soeiro A, Georgiev D, Jansen T, Gebel G, Bossard M, Christ M. Effect of a Strategy of Comprehensive Vasodilation vs Usual Care on Mortality and Heart Failure Rehospitalization Among Patients With Acute Heart Failure: The GALACTIC Randomized Clinical Trial. JAMA. 2019 Dec 17;322(23):2292-2302. doi: 10.1001/jama.2019.18598. PMID 31846016
- [Derived] Nyolczas N, Dekany M, Muk B, Szabo B. Combination of Hydralazine and Isosorbide-Dinitrate in the Treatment of Patients with Heart Failure with Reduced Ejection Fraction. Adv Exp Med Biol. 2018;1067:31-45. doi: 10.1007/5584_2017_112. PMID 29086392